CLINICAL TRIAL: NCT06435962
Title: Productive Value of Sonographic Measurement of Optic Nerve in Transitional Multiple
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Randa Alkady, resident doctor, Assiut University
Other Study IDs: optic nerve affection in RRMS
Record Dates: First submitted 2024-04-02; First posted 2024-05-30 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: sonography — measurement of optic nerve in RRMS by sonography and visual evoked potential( VEP) as correlation of axonal affection in RRMS patient
  Other Names: visual evoked potential( VEP)

SUMMARY:
1.to evaluate the potential role of the optic nerve diameter ( OND determined by ultrasonography and and visual nerve function by visual evoked potential as a biomarker of early axonal loss and disability in patients with relapsing remitting multiple sclerosis (RRMS).

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is one of the leading disabling neurological diseases in young Adults. Characteristically reliable biomarkers for every independent MS pathogenic factor are extremely important.

1 Increasing evidence has demonstrated that neuronal and axonal damage within the central nervous system (CNS) contributes substantially to the development of permanent disability in patients with MS

* 2 Thus, reliable, economic and easily assessable complementary surrogate biomarkers for axonal Degeneration and consequently disability remain to be identified
* 3 The optic nerve can serve as a useful clinical tool for studying these characteristics and can be used to Measure and monitor the pathological process of the disease. The optic nerve is most commonly assessed by ophthalmoscopy and magnetic resonance imaging (MRI), But measurement of the optic nerve diameter (OND) by a simple ultrasound examination and measurement of optic nerve function by visual evoked potential might permit a rough estimation of the extent of brain parenchymal involvement and the consequent global cerebral atrophy and disability In relapsing-remitting MS (RRMS) patients.

The analysis of the diameter of the optic nerve showed that it is possible To detect its atrophy in the affected eyes (with optic neuritis ) and, to a lesser extent, in un affected eye Also the visual evoked potential study has the ability to quantify the unsuspected clinically silent lesions, hence, allows confirming the vague deterioration of visual functions.

ELIGIBILITY:
1. inclusion criteria

   1. both sex
   2. Age group from 15 to 50 yrs
   3. Patient with RRMS without history of optic neuritis
2. Exclusion criteria :

   1. History of previous optic neuritis
   2. Medical illness of eye(e.g. diabetes and hypertension)
   3. MS patient on fingolimod for 6 months or more
   4. Relapsing or use of steroid in the past 3 months
   5. Proved alternative diagnosis (neuromyelitis optica )
   6. local eye disease or surgery

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: both sex and RRMS with out previous optic neuritis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
optic nerve measurement and correlation with axonal affection in RRMS | baseline
  measurement of optic nerve diameter and optic nerve sheath diameter (in millimeter) in predicting progression in RRMS (Relapsing remitting multiple sclerosis)

SECONDARY OUTCOMES:
2.Correlation of ultrasonography and visual evoked potential (change in p100 latency) with physical disability and cognitive score and fatigue by Multiple Sclerosis Functional Composite | Baseline
  Correlation of ultrasonography and visual evoked potential (change in p100 latency) with physical disability and cognitive score and fatigue by Multiple Sclerosis Functional Composite The score is based on a combination of timed tests of walking, arm function, and cognitive ability An integrated Multiple Sclerosis Functional Composite (MSFC) score is calculated using z-scores

CONTACTS AND LOCATIONS:
Overall Officials: Anwar M Ali, professor, Study Director — Assiut University

REFERENCES:
- [Background] Koraysha NA, Kishk N, Hassan A, Samy El Gendy NM, Shehata HS, Al-Azayem SA, Kamal YS. Evaluating optic nerve diameter as a possible biomarker for disability in patients with multiple sclerosis. Neuropsychiatr Dis Treat. 2019 Sep 6;15:2571-2578. doi: 10.2147/NDT.S216079. eCollection 2019. PMID 31564882
- [Background] De Masi R, Orlando S, Conte A, Pasca S, Scarpello R, Spagnolo P, Muscella A, De Donno A. Transbulbar B-Mode Sonography in Multiple Sclerosis: Clinical and Biological Relevance. Ultrasound Med Biol. 2016 Dec;42(12):3037-3042. doi: 10.1016/j.ultrasmedbio.2016.07.018. Epub 2016 Sep 15. PMID 27639433